CLINICAL TRIAL: NCT00160433
Title: A Phase II, 3-Month, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Three Doses of J867 (0.5, 1.5 and 5 mg QD) Versus Placebo in Subjects With Endometriosis
Brief Title: A Study to Evaluate the Safety and Effectiveness of Asoprisnil in the Treatment of Women With Endometriosis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Jenapharm GmbH & Co. KG (Unknown)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M01-398
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Endometriosis
Keywords: Pelvic pain; Dysmenorrhea; Dyspareunia; Infertility; asoprisnil
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Dysmenorrhea; Dyspareunia; Infertility | interventions — asoprisnil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil
- 2 (Experimental)
  Interventions: Drug: Asoprisnil
- 3 (Experimental)
  Interventions: Drug: Asoprisnil
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asoprisnil — 0.5 mg Tablet, oral Daily for 12 weeks
  Arms: 1
Drug: Asoprisnil — 1.5 mg Tablet, oral Daily for 12 weeks
  Arms: 2
Drug: Asoprisnil — 5.0 mg Tablet, oral Daily for 12 weeks
  Arms: 3
Drug: Placebo — Tablet, oral Daily for 12 weeks
  Arms: 4

SUMMARY:
The objective of this study is to determine the safety and efficacy of 3 asoprisnil doses (0.5 mg, 1.5 mg, and 5.0 mg) for 12 weeks in women with endometriosis.

DETAILED DESCRIPTION:
Endometriosis, the presence of endometrial tissue outside the uterus, is a progressive, estrogen-dependent disease that occurs in menstruating women of reproductive age. Although all major endometriosis therapies are effective for the treatment of pain, no single treatment is superior to others in terms of efficacy. The major drawbacks of the current medical therapies are severe side effects such as hot flushes and osteoporosis. The objective of this study is to determine if a dose-response relationship exists between asoprisnil and endometriosis-associated pelvic pain and dysmenorrhea or to establish the lowest effective dose of asoprisnil in the treatment of pelvic pain and dysmenorrhea associated with endometriosis. Women with surgically confirmed endometriosis will be administered asoprisnil 0.5, 1.5, and 5 mg tablets or a placebo once daily for 3 months and efficacy will be assessed by improvement in pelvic pain, dysmenorrhea, dyspareunia, bleeding, analgesic use, global efficacy, and quality of life questionnaires. Safety will be based on assessments of the endometrium, lipid profiles, adverse events, and changes from baseline laboratory values and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women (18-40 years)
* Surgically confirmed endometriosis within 3 years
* History of menstrual cycles between 21 and 35 days
* Moderate or severe pelvic pain OR moderate or severe dysmenorrhea OR moderate or severe pelvic tenderness accompanied by at least mild non-menstrual pelvic pain
* Negative pregnancy test
* Agrees to use double barrier method of contraception
* Pap smear with no evidence of malignancy or pre-malignant changes
* Ultrasound with no significant gynecological disorder.
* Otherwise in good health

Exclusion Criteria:

* Less than 3 months after having a baby or breast-feeding
* Any abnormal lab or procedure result the study-doctor considers important
* Severe reaction(s) to hormone therapy
* Anticipated need for excluded hormonal therapy or unapproved narcotics
* Current use of an IUD
* History or prolactinoma

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2002-08; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in pelvic pain as assessed by daily diary | Final month
Mean change from baseline in dysmenorrhea as assessed by daily diary | Final month

SECONDARY OUTCOMES:
Change from baseline in pelvic pain and dysmenorrhea scores from the daily diary. | Months 1,2,3 and Months 1-3
Change from baseline in dyspareunia and the combined pelvic pain/dysmenorrhea scores from the daily diary. | Months 1,2,3 and Months 1-3 and the Final Month
Change from baseline in the percentage of days with mild or greater combined pelvic pain/dysmenorrhea and moderate or greater combined pelvic pain/dysmenorrhea based on the daily diary. | Months 1,2,3 and Months 1-3 and Final Month
Change from baseline for pelvic pain, dysmenorrhea, dyspareunia, pelvic tenderness and induration scores assessed by the modified Biberoglu and Behrman pain scale. | Months 1,2,3 and Final Visit
Change from baseline in pelvic pain and dysmenorrhea assessed via the Visual Analog Scale. | Months 1,2,3 and Final Visit
Percent of subjects with "Yes" response to Global Efficacy question. | Months 1,2,3 and Final Visit
Change from baseline in analgesic use scores. | Months 1,2,3, Months 1-3 and Final Visit
Percent of subjects who achieve amenorrhea. | Throughout the treatment period
Change from baseline in Endometriosis Health Profile-30 (EHP-30) scores. | Month 3
Change from baseline in Short Form-36 scores. | Month 3
Change from baseline in both monthly bleeding scores and percentage of days with bleeding or spotting. | Months 1-3
Change from Screening menses in bleeding intensity. | First post-treatment menses
Change from baseline in hemoglobin and hematocrit. | Months 1,2,3 and Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott